CLINICAL TRIAL: NCT05518916
Title: Effects of Yakson Method Applied by Mother and Swaddling on Pain and Physiological Parameters During Heel Stick in Newborn
Brief Title: Effects of Yakson Method and Swaddling on Pain and Physiological Parameters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Aslihan Hacisalihoglu, Research Assistan, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IstanbulUC-AHacisalihoglu
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Pain During Heal Lancing
Keywords: nonfarmacology; pain; heal lancing; Yakson Method
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, three-arm randomized controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: After the researh report is written, a third person will assign an intervention and control group to the letters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yakson Method Group (Experimental): * The mother is informed about the benefits of the Yakson method.
  * Yakson method is taught practically to the mother. Education continues until the researcher is sure that the mother has done the method correctly. The mother starts the application 10 minutes before the heel lancing is done and continues for another 5 minutes after the heel lancing is done. During the application, the baby is recorded with the camera. Just before starting the Yakson method (initial assessment), at 10 minutes of the Yakson method (just before the heel lancing), during the heel lancing while the Yakson method is in progress, and 5 minutes after the procedure (just before the end of the tender touch), the newborn's pain and physiological parameters are evaluated. Evaluation results are recorded in the application observation form.
  Interventions: Other: Nonfarmacology method
- Swaddling Group (Experimental): * Parents are informed about the research and verbal consent is obtained.
  * Written consent is obtained with an informed consent form.
  * The Mother-Baby Information Form is filled.
  * Babies are fed 1 hour before blood collection.
  * And researher swaddling the baby
  Interventions: Other: Nonfarmacology method
- Control Group (No Intervention): Parents are informed about the research and verbal consent is obtained.
  * Written consent is obtained with an informed consent form.
  * The Mother-Baby Information Form is filled.
  * Babies are fed 1 hour before blood collection.
  * Before starting the heel lancing, a pulse oximeter probe will be attached to the baby's left big toe.
  * Blood is taken from the right heel of the foot.
  * During the application, the baby is recorded with the camera.
  * Evaluation results are recorded in the application observation form.

INTERVENTIONS:
Other: Nonfarmacology method — Yakson Method and Swaddling
  Arms: Swaddling Group; Yakson Method Group

SUMMARY:
Type of Study: The study was planned to be conducted in a randomized controlled experimental design.

Place and Time of the Research: Institutional permission will be obtained from the Balcalı Training and Research Hospital in Adana for the collection of research data. Researchers commit to start data collection after obtaining institutional permission. The data collection process will take 1 year after obtaining the institutional permission.

48 newborns who are suited the inclusion criteria will be included in the study. Participants will be assigned to 3 groups according to randomization: Swaddling, Yakson Method, and Control.

DETAILED DESCRIPTION:
Total processing time and baby's crying time are calculated by watching video recordings. In order to find the total procedure time, starting from the puncture of the baby's heel, the time until the dry cotton is placed on the baby's heel after the blood collection process is completed is calculated. The heart rate and SpO2 are noted by the investigator during the heel lancing procedure. Pain assessment of infants is done by two independent neonatal nurses, apart from the researcher, by watching video recordings. The scores given by the two observers will be evaluated by making inter-observer harmony. Before the evaluation, the nurses will be trained about the scale and its evaluation.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Newborn:

* Born at term (38-42 weeks)
* Healthy newborn
* Absence of congenital anomaly
* No analgesic or sedative medication has been administered in the last 6 hours
* Parent's consent for inclusion in the study in accordance with the consent form

Inclusion Criteria for Mother:

* Mother's willingness to participate in the study
* The mother can be mobilized and not have a physical disability (so that she can appyl Yakson therapy for her baby)
* Being communicative

Exclusion Criteria:

* Babies whose blood cannot be drawn on the first try

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Neonatal Infant Pain Scale (NIPS): | 1 year
  This scale was developed in 1993 by Lawrence et al. for premature and newborns. The scale measures the infant's response to pain behaviorally. The total score of the scale ranges from 0 to 7, and scores higher than 3 indicate the presence of pain.